CLINICAL TRIAL: NCT06512558
Title: Augmented Reality Feasibility for Non-invasive Preoperative Tracking in Breast Cancer Surgery
Acronym: AR-GBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02648-37
Record Dates: First submitted 2024-07-04; First posted 2024-07-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Subclinical Breast Cancer Lesion
MeSH Terms: interventions — Gadolinium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental)
  Interventions: Procedure: Additional MRI with gadolinium injection and 3D camera imaging

INTERVENTIONS:
Procedure: Additional MRI with gadolinium injection and 3D camera imaging — The study includes an additional MRI with gadolinium injection, performed in addition to standard practice. In addition, 3D camera images will be acquired at the time of surgery.

SUMMARY:
Breast cancer is diagnosed by imaging at a non-palpable stage in more than half of all cases. Surgical removal requires preoperative guidance. Generally, preoperative guidance is performed using a metal guide under local anaesthetic and radiological control. This type of guidance has several limitations. For the patient, it can be painful and traumatic. The procedure involves two departments: radiology and the operating theatre, which poses logistical constraints. What's more, between 10% and 40% of patients require repeat surgery for unhealthy margins, raising the question of the effectiveness of the tracking procedure. The investigators propose to develop a non-invasive intraoperative guidance system: Augmented Reality, which will provide a 3D vision with virtual transparency of the breast during surgery, thanks to real-time fusion of preoperative imaging with video from a camera located in the operating room. The process is illustrated below.

Illustration of the general principle of the augmented reality system for locating non-palpable breast lesions. The images above represent a preliminary test carried out on the computer outside the operating room. This is an initial research prototype which has not yet been validated and is not suitable for routine use.

ELIGIBILITY:
Inclusion Criteria:

* Major women
* Requiring conservative surgical management of a subclinical cancerous breast lesion (not palpable), the histology of which has been previously proven by anatomopathology;
* Having a breast MRI indication at the time of the breast assessment performed at the Centre Jean Perrin
* Ability to give informed consent to participate in the study,
* Membership of a social security scheme

Exclusion Criteria:

* Patients with breast neoplasia during pregnancy;
* Persons deprived of their liberty or under guardianship or incapable of giving consent;
* Refusal to participate.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the study | 1 year
  The feasibility of the study will be considered to have been achieved if the investigators obtain at least 4 successes among the 5 patients who benefited from the augmented reality procedure pre- and intraoperatively.
  Success is defined at both preoperative and intraoperative levels. Success in the preoperative phase is defined by: visibility of registration landmarks (clavicle, sternal fork, sternum, xyphoid process and areolar-nipple plate).
  Success in the intraoperative phase is defined by: non-prolongation of anesthesia time due to the study procedure.

SECONDARY OUTCOMES:
Time measurement of the study procedure | 1 year
  Measurement of the time required to complete the various stages of the study procedure and surgery : device set-up, marking of registration marks on the patient's bust with a dermographic pencil, 3D acquisition of the patient's bust using a 3D camera, duration of the procedure, anesthesia time.
Creating a phantom | 1 year
  Success of creating a phantom is deemed to have been achieved if the breast Phantom including all clinical features
Assessment of the feasibility of images fusion | 1 year
  Assessment of the feasibility of fusing supine 3D breast MRI images and post-MRI ultrasound (second look) with target lesion detection.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Jean PERRIN, Clermont-Ferrand, France